CLINICAL TRIAL: NCT06982131
Title: A Phase I, Randomized, Investigator/Participant-Blind, Placebo-Controlled, Fixed-Sequence Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of Orally Administered RO7795081 and the Effect of Steady-State Dose of Orally Administered RO7795081 on the Pharmacokinetics of Pitavastatin and Rosuvastatin in Otherwise Healthy Overweight or Obese Adult Participants
Brief Title: A Study Investigating the Safety of RO7795081 and the Effect of RO7795081 on How the Body Processes Pitavastatin and Rosuvastatin in Otherwise Healthy Overweight or Obese Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BP45800; 2024-519277-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Rosuvastatin Calcium; pitavastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: ROS Alone, Then PIT Alone, Then RO7795081 Alone, Then RO7795081 + ROS, Then RO7795081 + PIT (Experimental): Period 1: Rosuvastatin (ROS) alone; Period 2: Pitavastatin (PIT) alone; Period 3: RO7795081 alone; Period 4: RO7795081 in combination with ROS; Period 5: RO7795081 in combination with PIT
  Interventions: Drug: RO7795081; Drug: Rosuvastatin; Drug: Pitavastatin
- Arm 2: ROS Alone, Then PIT Alone, Then Placebo Alone, Then Placebo + ROS, Then Placebo + PIT (Placebo Comparator): Period 1: Rosuvastatin (ROS) alone; Period 2: Pitavastatin (PIT) alone; Period 3: Placebo alone; Period 4: Placebo in combination with ROS; Period 5: Placebo in combination with PIT
  Interventions: Drug: Placebo; Drug: Rosuvastatin; Drug: Pitavastatin

INTERVENTIONS:
Drug: RO7795081 — RO7795081 will be administered orally during Periods 3, 4, and 5, according to the protocol.
  Other Names: CT-996; RG6652
  Arms: Arm 1: ROS Alone, Then PIT Alone, Then RO7795081 Alone, Then RO7795081 + ROS, Then RO7795081 + PIT
Drug: Placebo — Placebo will be administered orally during Periods 3, 4, and 5, according to the protocol.
  Arms: Arm 2: ROS Alone, Then PIT Alone, Then Placebo Alone, Then Placebo + ROS, Then Placebo + PIT
Drug: Rosuvastatin — A single 10 mg dose of rosuvastatin (ROS) will be taken on Day 1 of Period 1 and on Day 1 of Period 4.
  Other Names: Crestor®
Drug: Pitavastatin — A single 1 mg dose of pitavastatin (PIT) will be taken on Day 1 of Period 2 and on Day 1 of Period 5.
  Other Names: Livazo®; Livalo®; Zypitamag®

SUMMARY:
This is a randomized, investigator-and-participant-blind, placebo-controlled, fixed sequence, cross-over, Phase 1 study to investigate the safety, tolerability, and pharmacokinetics of multiple doses of orally administered RO7795081 and the effect of a steady-state dose of orally administered RO7795081 on the pharmacokinetics of pitavastatin and rosuvastatin in otherwise healthy, overweight or obese adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with no clinically relevant findings on physical examination at screening and at baseline (including detailed medical and surgical history, vital signs, 12-lead ECG, hematology, blood chemistry, and urinalysis); with no suspicion of cognitive impairment or dementia as judged by the Investigator; who are not under judicial supervision, guardianship, or curatorship.
* Body Mass Index (BMI) ≥27.0 kg/m^2 at screening and on Day -1 of Period 1
* Stable body weight (defined as <5% gain or loss) in the 2 months prior to screening as per verbal report by the participant and for the period between screening and Day -1 of Period 1 as per measured weight
* Agreement to adhere to the contraception requirements

Exclusion Criteria:

* Pregnant, breastfeeding, or intending to become pregnant during the study
* Any condition or disease detected during the medical interview or physical examination that would render the participant unsuitable for the study, place the participant at undue risk, or interfere with the ability of the participant to complete the study in the opinion of the Investigator
* History or presence of any clinically significant cardiovascular, broncho-pulmonary, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological, psychiatric, or metabolic disorders, allergic diseases, hypofertility, cancer, or cirrhosis
* History or evidence of any medical condition capable of significantly altering the absorption, metabolism, or elimination of drugs
* History of convulsions (other than benign febrile convulsions of childhood) including epilepsy, or personal history of significant cerebral trauma or CNS infections (e.g., meningitis)
* History of acute or chronic metabolic acidosis, including diabetic ketoacidosis with or without coma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | From the first dose of study treatment until the final visit (up to 111 days)
Incidence of Abnormal Clinical Laboratory Test Results | From the first dose of study treatment until the final visit (up to 111 days)
Incidence of Abnormal Vital Sign Assessments | From the first dose of study treatment until the final visit (up to 111 days)
Incidence of Abnormal Electrocardiogram Parameters | From the first dose of study treatment until the final visit (up to 111 days)
Maximum Plasma Concentration Observed (Cmax) of Rosuvastatin, Administered Alone and in Combination with RO7795081 | Periods 1 and 4: predose and postdose at prespecified times on Days 1 to 5
Time to Maximum Plasma Concentration (Tmax) of Rosuvastatin, Administered Alone and in Combination with RO7795081 | Periods 1 and 4: predose and postdose at prespecified times on Days 1 to 5
Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to the Last Measurable Concentration (AUClast) of Rosuvastatin, Administered Alone and in Combination with RO7795081 | Periods 1 and 4: predose and postdose at prespecified times on Days 1 to 5
AUC from Time 0 to Infinity (AUCinf) of Rosuvastatin, Administered Alone and in Combination with RO7795081 | Periods 1 and 4: predose and postdose at prespecified times on Days 1 to 5
Cmax of Pitavastatin, Administered Alone and in Combination with RO7795081 | Periods 2 and 5: predose and postdose at prespecified times on Days 1 to 4
Tmax of Pitavastatin, Administered Alone and in Combination with RO7795081 | Periods 2 and 5: predose and postdose at prespecified times on Days 1 to 4
AUClast of Pitavastatin, Administered Alone and in Combination with RO7795081 | Periods 2 and 5: predose and postdose at prespecified times on Days 1 to 4
AUCinf of Pitavastatin, Administered Alone and in Combination with RO7795081 | Periods 2 and 5: predose and postdose at prespecified times on Days 1 to 4

SECONDARY OUTCOMES:
Plasma Concentration of RO7795081 Over Time, Administered Alone and in Combination with Rosuvastatin and Pitavastatin | Period 3: predose and postdose at prespecified times from Days 2 to 49; Period 4: predose and postdose at prespecified times on Days 1 to 4; Periods 4: predose and postdose at prespecified times on Days 1 to 9
Cmax of RO7795081, Administered Alone and in Combination with Rosuvastatin and Pitavastatin | Period 3: predose and postdose at prespecified times from Days 2 to 49; Period 4: predose and postdose at prespecified times on Days 1 to 4; Periods 4: predose and postdose at prespecified times on Days 1 to 9
Tmax of RO7795081, Administered Alone and in Combination with Rosuvastatin and Pitavastatin | Period 3: predose and postdose at prespecified times from Days 2 to 49; Period 4: predose and postdose at prespecified times on Days 1 to 4; Periods 4: predose and postdose at prespecified times on Days 1 to 9
AUClast of RO7795081, Administered Alone and in Combination with Rosuvastatin and Pitavastatin | Period 3: predose and postdose at prespecified times from Days 2 to 49; Period 4: predose and postdose at prespecified times on Days 1 to 4; Periods 4: predose and postdose at prespecified times on Days 1 to 9
AUCinf of RO7795081, Administered Alone and in Combination with Rosuvastatin and Pitavastatin | Period 3: predose and postdose at prespecified times from Days 2 to 49; Period 4: predose and postdose at prespecified times on Days 1 to 4; Periods 4: predose and postdose at prespecified times on Days 1 to 9

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- ICON Plc (LPRA) - Netherlands, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No